CLINICAL TRIAL: NCT01001026
Title: PCIRN Evaluation of Pandemic H1N12009 Influenza Vaccine in Aboriginal Children and Adults
Brief Title: Rapid Evaluation of Pandemic H1N1 Influenza Vaccine in Aboriginal Children and Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Scheifele (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Sponsor-Investigator, David Scheifele, Principal Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H09-02769
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: H1N1/2009 Influenza
Keywords: vaccine; H1N1; influenza; H1N1 influenza vaccine; pandemic
MeSH Terms: conditions — Influenza, Human | interventions — arepanrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Adults: One doses of H1N12009 vaccine
  Interventions: Biological: Arepanrix
- 2 (Other): Children: Two doses of H1N12009 vaccine given 3 weeks apart
  Interventions: Biological: Arepanrix

INTERVENTIONS:
Biological: Arepanrix — Adults: One dose Arepanrix vaccine given IM (0.5 mL)
  Arms: 1
Biological: Arepanrix — Children: Two doses of Arepanrix vaccine given IM (0.25 mL) three weeks apart
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety and effectiveness (immune response) to a licensed H1N12009 influenza vaccine in aboriginal children and adults. The study will enroll 200 healthy adults (ages 20-59 years) and 75 healthy children (ages 6-35 months). Adults will receive one dose of a licensed H1N1 vaccine and children will receive two doses of a licensed H1N1 vaccine approximately 3 weeks apart. Study procedures include: medical history, blood samples and completing a memory aid. Participants will be involved in study related procedures for approximately 3 weeks (adults) or 6 weeks (children).

DETAILED DESCRIPTION:
During the first wave of the H1N12009 pandemic in Canada, persons of aboriginal background were more often hospitalized with severe infections than were other Canadians. Among First Nations members the hospitalization rate was 5 times higher than the national average. Common risk factors were young age (children and younger adults) and underlying health conditions. A high proportion of aboriginal adults have health conditions that predispose to adverse influenza outcomes, including diabetes, asthma, obesity and smoking-related lung diseases.

Aboriginals could benefit substantially from timely, effective vaccination against pandemic influenza and are expected to be among the first Canadians to be offered vaccine when available. The vaccine dosing recommendation will be based on limited studies in the general population, leaving open the question of whether aboriginals will respond satisfactorily to the recommended dosing. Unique social and biological factors among aboriginals could affect their responses to vaccination, reducing protection or increasing adverse effects. Thus it would be optimal to evaluate the safety and immunogenicity of the pandemic vaccine among the earliest aboriginal recipients, to inform the subsequent vaccination of other aboriginal groups.

The objectives of this study are two-fold:

1. To evaluate the safety and immunogenicity of H1N12009 influenza vaccine in a convenience sample of children and adults of aboriginal background (First Nations, Metis and Inuit) with emphasis on subgroups at greatest risk of severe disease.
2. To complete this evaluation soon after the pandemic vaccines become available so as to inform the subsequent use of the vaccines in the aboriginal population.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Written informed consent provided by or for the subject
* Aboriginal ethnicity (First Nations, Metis or Inuit)
* Adults 20-59 years of age
* Children 6-35 months of age

Exclusion Criteria:

* Allergies to eggs, thimerosal or gentamicin sulphate
* Life-threatening reaction to previous Flu vaccine
* Bleeding disorder
* Pregnancy
* Receipt of blood or blood products in past 3 months
* Compromised immune system
* Chronic illness
* Previous lab-confirmed H1N1/2009 infection

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) for days 0-6 after each vaccination | Day 7 and Day 21 post vaccination
Occurrence of serious adverse events (SAEs) and other significant health events up to 21 days after each vaccination | Day 7 and Day 21 post vaccination

SECONDARY OUTCOMES:
Comparison of baseline and post-immunization antibody titres | Day 21 (adults) and Day 42 (children)

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, MD, Principal Investigator — University of British Columbia; Ethan Rubinstein, MD, Study Director — University of Manitoba Health Sciences Centre; Gerald Predy, MD, Study Director — Alberta Health Services, Edmonton; Laura Sauve, MD, Study Director — University of British Columbia
Locations (5):
- Canada (5):
  - Calgary Health Services and Alberta Children's Hospital, Calgary, Alberta
  - Capital Health District, Alberta Health Services, Edmonton, Alberta
  - Child and Family Research Center, Vancouver, British Columbia
  - Vaccine Evaluation Center, University of British Columbia, Vancouver, British Columbia
  - University of Manitoba Health Sciences Centre, Winnipeg, Manitoba

REFERENCES:
- [Derived] Rubinstein E, Predy G, Sauve L, Hammond GW, Aoki F, Sikora C, Li Y, Law B, Halperin S, Scheifele D. The responses of Aboriginal Canadians to adjuvanted pandemic (H1N1) 2009 influenza vaccine. CMAJ. 2011 Sep 20;183(13):E1033-7. doi: 10.1503/cmaj.110196. Epub 2011 Jul 25. PMID 21788422